CLINICAL TRIAL: NCT02673294
Title: Chronicity Dependence of a Balance Training in Adults Post-stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospitales Nisa (Other)
Collaborators: Universitat Politècnica de València (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HNISA2016-01
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Stroke, Postural Balance, Virtual Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- intervention (6-12 months) (Experimental): Participants with a chronicity between 6-12 months
  Interventions: Other: balance virtual rehabilitation
- Intervention (12-24 months) (Experimental): Participants with a chronicity between 12-24 months
  Interventions: Other: balance virtual rehabilitation
- Intervention (>24 months) (Experimental): Participants with a chronicity >24 months
  Interventions: Other: balance virtual rehabilitation

INTERVENTIONS:
Other: balance virtual rehabilitation

SUMMARY:
The level of stroke chronicity has been proposed as an influential variable related to functional balance. However, little is known about the effect of this variable on the effectiveness and maintenance of gains of physical therapy interventions on balance. The objective of this study is to determine the influence of time since injury on the rehabilitation of balance after stroke. Participants will be assigned to a least (6-12 months), a moderate (12-24 months), or a most chronic (> 24 months) group. All the participants will train for 20 one-hour sessions, administered three to five times a week, combining conventional physical therapy exercises and customized exercises interfaced on a balance board that promotes the training of the ankle and hip strategies. Participants will be assessed before, after the intervention, and one month later with a posturography test (sway speed and limits of stability) and clinical scales (Berg Balance Scale, Functional Reaches Test, 30-Second Sit-to-Stand Test, Timed Up and Down Stairs Test, Stepping Test, Timed Up-and-Go Test, and the 10-meter Walking Test).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 and ≤ 65 years old
* Chronicity > six months
* Fairly good cognitive condition defined by scores in the Mini-Mental State Examination above 23
* Ability to walk 10 meters indoors with or without technical orthopaedic aids.

Exclusion Criteria:

* Impaired comprehension that hinder sufficient understanding of the instructions defined by Mississippi Aphasia Screening Test scores below 45
* Unilateral spatial neglect
* Ataxia or any other cerebellar symptom
* Severe auditory or visual impairments
* Motional or behavioural circumstances that impede adequate collaboration.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-02; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Balance Berg Scale | up to 1-month follow-up